CLINICAL TRIAL: NCT03163030
Title: Autonomic Neural Regulation Therapy to Enhance Myocardial Function in Heart Failure With Preserved Ejection Fraction (ANTHEM-HFpEF) Study
Brief Title: Autonomic Regulation Therapy in Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Organization: LivaNova (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-04
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure; Preserved Ejection Fraction; VNS; Vagus Nerve; Autonomic Regulation Therapy
MeSH Terms: conditions — Heart Failure | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy (Experimental): Right Cervical Vagus Nerve Stimulation (VNS)
  Interventions: Device: Vagus Nerve Stimulation (VNS)

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS) — Electrical Stimulation of the Vagus Nerve

SUMMARY:
The ANTHEM-HFpEF Study is designed to demonstrate the safety and efficacy of vagus nerve stimulation (VNS) with the Cyberonics VNS Therapy System for the treatment of subjects with symptomatic heart failure with preserved and mid-range ejection fraction.

DETAILED DESCRIPTION:
Heart failure patients will be enrolled and implanted with a cervical VNS system on the right side. After a 2-week post-implantation recovery period and a 10-week stimulation titration period, continuous periodic stimulation will be performed for 12 months, with data collection at 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic heart failure, New York Heart Association (NYHA) class II/III with preserved and mid-range EF (≥40%).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 12 months
  Incidence of procedure and device-related complications

SECONDARY OUTCOMES:
Cardiac Size (LAVI) | 12 months
  Left atrial volume index
Functional Status (6MWD) | 12 months
  6-minute walk distance
Quality of Life Score | 12 months
  Minnesota Living with Heart Failure Questionnaire score
Functional Status (NYHA Class) | 12 months
  New York Heart Association classification
Cardiac Function (E/E') | 12 months
  Ratio of mitral velocity to early diastolic velocity of the mitral annulus
Cardiac Size (LV mass index) | 12 months
  Left ventricular mass index
Autonomic Function (HRV) | 12 months
  Heart rate variability
Blood Biomarkers | 12 months
  Blood Levels of Heart Failure Biomarkers (NT-proBNP, creatinine, C-reactive protein)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Libbus, Ph.D, Study Director — Cyberonics, Inc.
Locations (1):
- Krishna Institute of Medical Science, Secunderabad, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kumar HU, Nearing BD, Mittal S, Premchand RK, Libbus I, DiCarlo LA, Amurthur B, KenKnight BH, Anand IS, Verrier RL. Autonomic regulation therapy in chronic heart failure with preserved/mildly reduced ejection fraction: ANTHEM-HFpEF study results. Int J Cardiol. 2023 Jun 15;381:37-44. doi: 10.1016/j.ijcard.2023.03.030. Epub 2023 Mar 17. PMID 36934987